CLINICAL TRIAL: NCT00183378
Title: Behavioral Treatment of Nocturnal Disturbances in Alzheimer's Disease
Brief Title: Using Behavioral Programs to Treat Sleep Problems in Individuals With Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sue McCurry, Research Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH072736 (NIH); R01MH072736 (NIH); DATR A4-GPS
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Alzheimer Disease; Sleep Initiation and Maintenance Disorders
Keywords: Alzheimer's Disease; Insomnia; Sleep Problems; Elderly; Caregivers
MeSH Terms: conditions — Alzheimer Disease; Sleep Initiation and Maintenance Disorders; Parasomnias | interventions — Walking; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Routine medical care with education: therapist provides information about the nature of sleep changes in people with Alzheimer's disease, general information about treatments for insomnia, and caregiver support.
  Interventions: Behavioral: Routine Medical Care with Education
- 2 (Active Comparator): Walking: the therapist introduces a walking program and assists the caregiver in establishing a daily walking routine of 30 minutes for the study participant.
  Interventions: Behavioral: Walking Program
- 3 (Active Comparator): Light exposure: the therapist provides a light box and teaches the caregiver how to use the box so that the study participant's daily exposure to bright light is one hour.
  Interventions: Behavioral: Light Exposure Program
- 4 (Active Comparator): Combination: the therapist provides education plus assistance setting up an individualized sleep program, a daily walking routine, and a schedule for daily light exposure.
  Interventions: Behavioral: Combined Education, Walking and Light Exposure Program

INTERVENTIONS:
Behavioral: Walking Program — The therapist introduces a walking program and assists the caregiver in establishing a walking routine of 30 minutes/day for the study participant.
  Arms: 2
Behavioral: Light Exposure Program — The therapist provides a light box and teaches the caregiver how to use the box so that the study participant's daily exposure to bright light is one hour.
  Arms: 3
Behavioral: Combined Education, Walking and Light Exposure Program — The therapist provides a combination of education plus assistance setting up an individualized sleep program, a daily walking routine, and a schedule for daily light exposure.
  Arms: 4
Behavioral: Routine Medical Care with Education — The therapist provides information about the nature of sleep changes in people with Alzheimer's disease, general information about treatments for insomnia, and caregiver support. Participants are free to use whatever medical services they wish during study participation.
  Arms: 1

SUMMARY:
This study will compare four different behavioral treatment programs to determine which is most effective in reducing night-time disturbances in individuals with Alzheimer's disease (AD).

DETAILED DESCRIPTION:
Nocturnal disturbances, such as getting out of bed repeatedly, having hallucinations, talking or singing in bed, and waking up confused are common among patients with AD. Such nocturnal disturbances are associated with increased physical and psychological morbidity in both AD patients and their caregivers and are a major risk factor for patient institutionalization. Nonpharmacologic treatments for these disturbances are needed. This study will assign AD patients to one of four different treatments to determine which is most effective in reducing nocturnal disturbances.

This study will last 6 months. Participants will be randomly assigned to a walking program, a light exposure program, a "NITE-AD" program, combining the walking and light exposure programs, or routine AD care with nocturnal disturbance education. Walking program participants will have three 1-hour visits with a therapist over an 8-week period. The therapist and the participant will set an initial daily walking goal and develop a plan for gradually increasing the participants' walking to 30 minutes/day, to be increased at a participant-selected pace. Pedometers will be given to participants to monitor daily activity. The therapist will also discuss exercise safety and will review ways to prevent muscle soreness. Light program participants will also have three 1-hour visits with a therapist over 8 weeks. The therapist will develop a daily, caregiver-supervised light exposure plan requiring participants to sit in front of a light box for 1 hour every day. NITE-AD program participants will have six 1-hour visits with a therapist over 8 weeks; their visits will include setting up both walking and the light exposure routines. Participants assigned to education will receive information about about sleep in aging and dementia, but no assistance setting up walking or light exposure plans.

Participants will be assessed at study entry and at Months 2 (post-test) and 6. The sleep patterns of both the patients and the caregivers will be measured. Caregiver reports of patients' night-time behavioral disturbances and readings from an actigraph, a small electronic device worn by participants that records and reports their levels of activity at night, will be used to estimate sleep. The study will also collect data on patient and caregiver mood, stress, and behavior. A follow-up visit will occur 6 months after study completion; at the follow-up visit, the same outcome measures will be collected as at baseline and post-test. Participants will receive 3 biannual phone follow-ups (12, 18, and 24 months) to assess patient residential status and caregiver reports of patient and caregiver sleep.

ELIGIBILITY:
Inclusion Criteria for Alzheimer's Disease Patients:

* Diagnosis of probable or possible Alzheimer's Disease
* Have at least two sleep disturbances, occurring 3 or more times per week
* Reside in a residential home with a family member caregiver
* Able to walk without assistance

Exclusion Criteria for Alzheimer's Disease Patients:

* Pre-existing diagnosis of a primary sleep disorder, such as sleep apnea or periodic limb movement disorder
* Blindness
* Current use of photosensitizing medication

Inclusion Criteria for Family Caregiver:

* Currently caring for a family member with Alzheimer's disease

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2005-09; Primary Completion 2009-09 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Patient total wake time (actigraphy) | Measured 3 times over 6 months
Caregiver reports of patient behavioral disturbances at night (Sleep Disorders Inventory) | Measured 3 times over 6 months

SECONDARY OUTCOMES:
Additional patient actigraphy outcomes | Measured 3 times over 6 months
Patient daytime sleepiness, behavioral problems, and residential status | Measured 3 times over 6 months
Caregiver sleep | Measured 3 times over 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan M. McCurry, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] McCurry SM, Gibbons LE, Logsdon RG, Vitiello M, Teri L. Training caregivers to change the sleep hygiene practices of patients with dementia: the NITE-AD project. J Am Geriatr Soc. 2003 Oct;51(10):1455-60. doi: 10.1046/j.1532-5415.2003.51466.x. PMID 14511168
- [Background] McCurry SM, Gibbons LE, Logsdon RG, Vitiello MV, Teri L. Nighttime insomnia treatment and education for Alzheimer's disease: a randomized, controlled trial. J Am Geriatr Soc. 2005 May;53(5):793-802. doi: 10.1111/j.1532-5415.2005.53252.x. PMID 15877554
- [Result] McCurry SM, Pike KC, Logsdon RG, Vitiello MV, Larson EB, Teri L. Predictors of short- and long-term adherence to a daily walking program in persons with Alzheimer's disease. Am J Alzheimers Dis Other Demen. 2010 Sep;25(6):505-12. doi: 10.1177/1533317510376173. Epub 2010 Jul 26. PMID 20660515
- [Result] McCurry SM, Pike KC, Vitiello MV, Logsdon RG, Larson EB, Teri L. Increasing walking and bright light exposure to improve sleep in community-dwelling persons with Alzheimer's disease: results of a randomized, controlled trial. J Am Geriatr Soc. 2011 Aug;59(8):1393-402. doi: 10.1111/j.1532-5415.2011.03519.x. Epub 2011 Jul 28. PMID 21797835